CLINICAL TRIAL: NCT06776029
Title: A Prospective, Single-Arm Trial of Fecal Microbiota Transplantation for Hemorrhagic Radiation-Induced Rectal Injury
Brief Title: Fecal Microbiota Transplantation for Radiation-Induced Proctopathy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRP202401
Record Dates: First submitted 2025-01-10; First posted 2025-01-15 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Radiation Induced Proctitis
Keywords: fecal microbiota transplantation; rectal bleeding; radiation proctitis
MeSH Terms: conditions — Gastrointestinal Hemorrhage | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Fecal Microbiota Transplantation (Experimental): Fecal microbiota capsules are given by 8 sessions over a 12-week period, with the initial 3 sessions every other day in the first week and the subsequent sessions every two weeks. The FMT regimen involves oral intake of 40 capsules per session. The best supportive care is performed when necessary, including oral medicine, enema, blood transfusion, and endoscopic procedures.
  Interventions: Biological: Fecal Microbiota Transplantation Capsule

INTERVENTIONS:
Biological: Fecal Microbiota Transplantation Capsule — FMT is delivered via oral capsules. Fecal microbiota capsules are given by 8 sessions over a 12-week period, with the initial 3 sessions every other day in the first week and the subsequent sessions every two weeks. The FMT regimen involves oral intake of 40 capsules per session. The best supportive care is performed when necessary, including oral medicine, enema, blood transfusion, and endoscopic procedures.

SUMMARY:
The goal of this single-arm trial is to learn if Fecal Microbiota Transplantation (FMT) works to treat hemorrhagic radiation-induced proctopathy. The main questions it aims to answer are:

* Dose FMT alleviate the symptom of severe rectal bleeding?
* Dose FMT improve the endoscopic findings of proctopathy?

Participants will:

* Take fecal microbiota capsules by 8 sessions over a 12-week period.
* Visit the clinic once every 4 weeks for checkups and tests.
* Keep a diary of their symptoms and the number of times they use other supportive care.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-75 years old
* At least 3 months since the completion of pelvic radiotherapy
* No evidence of tumor recurrence or metastasis
* Rectal bleeding with grade 2-4 by LENT-SOMA scales
* Colonoscopy indicating rectal congested mucosa or telangiectasia
* Poor response to supportive care, or hemoglobin level less than or equal to 70 g/L in the past 3 months

Exclusion Criteria:

* Acute or chronic infectious diseases
* Serious systemic diseases
* Known allergies to any components of the study medication
* Colonoscopy indicating rectal ulceration (>1cm2), fistula, stricture, or necrosis
* Late complications related to pelvic radiation injury
* Other hemorrhagic or coagulation disorders
* Previous rectal resection
* Bowel obstruction or perforation that require surgery
* Cognitive or psychological disorder
* Contraindications to FMT administration

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with mild rectal bleeding (grade 0-1) | At the time of 12 weeks since the start of treatment
  The symptom of rectal bleeding will be assessed by LENT-SOMA scales

SECONDARY OUTCOMES:
Number of participants with mild rectal bleeding (grade 0-1) | At the time of 24 weeks since the start of treatment
  The symptom of rectal bleeding will be assessed by LENT-SOMA scales
Number of participants with improved colonoscopic findings | At the time of 12 and 24 weeks since the start of treatment
  The colonoscopic findings will be assessed by the Vienna Rectoscopy Score.

CONTACTS AND LOCATIONS:
Locations (1):
- The Sixth Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No